CLINICAL TRIAL: NCT04840355
Title: Clinical Study on Multidimensional Prevention of Sintilimab Induced irAEs Based on GEP Pattern Recognition
Brief Title: Multi-Centre, Prospective, Non-Interventional Study to Intensively Monitor the Safety of Sintilimab in Clinical Practice Among Chinese Patients
Status: Recruiting | Type: Observational
Sponsor: Guohui Li (Other)
Responsible Party: Sponsor-Investigator, Guohui Li, Head of Pharmacy department, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Organization: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Other Study IDs: LC2020L03
Record Dates: First submitted 2021-04-07; First posted 2021-04-12 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Immune Related Adverse Events; PD-1
MeSH Terms: interventions — sintilimab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Subjects with no irAEs
  Interventions: Drug: Sintilimab Injection
- Subjects with degree 1-2 irAEs
  Interventions: Drug: Sintilimab Injection
- Subjects with degree 3-4 irAEs
  Interventions: Drug: Sintilimab Injection

INTERVENTIONS:
Drug: Sintilimab Injection — The recommended dose for intravenous infusion is 200 mg on day 1.Courses repeat every 21 days for up to 6 months in the absence of disease progression or unacceptable toxicity.

SUMMARY:
In recent years, immunotherapy has become one of the important treatments for malignant tumors. Among them, PD-1 inhibitors have been widely used in clinical practice, and have shown a significant survival benefits in many patients. However, the incidence of immune-related adverse reactions (irAEs) of PD-1 inhibitors is relatively high, and severe cases can even threaten patients's life. At present, irAEs have become a bottleneck and it is urgent to establish a prevention strategy for the prediction of irAEs. In this study, the investigators intends to use Sintilimab as the research drug. A prospective cohort study was carried out. Part of the sample which was used as a training set would be detected for producing a time-series multi-dimensional data such as differential genes, metabolites and immune factors. Then gene expression programming (GEP) was used to explore the irAEs recognition model. Then, based on this recognition model, internal verification ( part of samples from the center 1 ) and external verification ( part of samples from the center 2 and center 3 samples) are carried out to accurately predict the high-risk population of irAEs and realize the early-stage warning of Sintilimab induced- irAEs.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 and ≤75 years old;
2. Subjects with histologically or cytologically confirmed are prepared to receive Sintilimab treatment;
3. Life expectancy of at least 6 months;
4. Eastern Cooperative Oncology Group (ECOG) PS status≤ 2 or Karnofsky (KPS) ≥ 60;
5. No prior immune checkpoint inhibitor treatment
6. Signed written informed consent before any study-related procedure;
7. Adequate hematopoietic function as defined by an absolute neutrophil count ≥1.5×109 /L, platelet count≥80×109 /L, hemoglobin≥90 g/L
8. Adequate hepatic function, defined as a total bilirubin level≤1.5 ×upper limit of normal (ULN); aspartate aminotransferase (AST) and alanine aminotransferase (ALT) levels ≤2.5 × ULN in subjects without liver metastases, AST and ALT levels ≤5 × ULN in subjects with documented liver metastases;
9. Adequate renal function, defined as serum creatinine (Cr)≤1.5×ULN or calculated creatinine clearance≥60ml/min (Cockcroft-Gault formula);
10. Serum albumin ≥28g/L;
11. Thyroid-stimulating hormone (TSH)≤1×ULN (if abnormal,subject with the normal levels of FT3 and FT4 can be enrolled).

Exclusion Criteria:

1. Has active autoimmune disease;
2. Severe heart, lung, brain, kidney, gastrointestinal or systemic diseases;
3. has interstitial lung disease;
4. Simultaneous use of drugs that can affect the results of this study;
5. Treatment may interfere with the results of the study
6. Allergy or intolerance to the study drug
7. subject with unconsciousness and psychiatric disorder
8. Pregnant and lactating women
9. Subject with poison and alcohol abuse

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with histologically or cytologically confirmed are prepared to receive Sintilimab treatment
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-02-26 (Actual); Primary Completion 2025-11-14 (Estimated); Study Completion 2025-11-14 (Estimated)

PRIMARY OUTCOMES:
irAEs | 24 month
  degree of irAEs induced by Sintilimab Injection

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided